CLINICAL TRIAL: NCT01703923
Title: An Exploratory, Randomized, Placebo-Controlled, Double-Blind, Crossover Study of FP01 Lozenges in Subjects With Chronic Refractory Cough
Brief Title: An Exploratory Study of FP01 Lozenges in Subjects With Chronic Refractory Cough
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avalo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Clin01-003
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Refractory Cough

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FP01 6mg or Placebo (Experimental): FP01 6mg Oral
  Interventions: Drug: FP01; Drug: placebo
- FP01 12mg or Placebo (Experimental): FP01 12mg Oral
  Interventions: Drug: FP01; Drug: placebo

INTERVENTIONS:
Drug: FP01
Drug: placebo

SUMMARY:
The purpose of this study is to determine the antitussive effect size and dose response of FP01 lozenges in subjects with chronic cough and to demonstrate the safety and tolerability of FP01 lozenges in subjects with chronic cough.

ELIGIBILITY:
Inclusion Criteria:

* Subject must sign an Institutional Review Board approved informed consent and agree to complete required clinic visits
* Subjects must be able to read and write English
* Subject must exceed a cough severity threshold (VAS) during screening visit (Cough Severity VAS Score ≥ 35 mm)
* Mean CSD frequency domain (Only Questions 1-3 at time of screening) score > 3.0
* Stable chest X-ray
* Forced expiratory volume 1 (FEV1) and forced vital capacity (FVC) >70% predicted measured using spirometry
* Body mass index (BMI) 18.5 - 38
* Subjects must be non-smokers or have refrained from using nicotine or nicotine containing products for at least 6 months
* Female subjects should be either post-menopausal (amenorrhea for at least 12 consecutive months), surgically sterile, or women of child-bearing potential with a negative serum beta human chorionic gonadotropin pregnancy test prior to entering the study and who are using or agree to use an acceptable method of contraception as determined by the Investigator

Exclusion Criteria:

* Recent significant change in pulmonary status or upper respiratory tract infection (<4 weeks of randomization)
* Female subjects who are pregnant, breast feeding or sexually active without contraception.
* History of chronic obstructive pulmonary disease (COPD)
* History of asthma that required any significant change in treatment within 2 weeks of randomization. Subjects with asthma are eligible as long as the subject is not being treated with oral steroids but may enroll as long as no new medication to control their asthma has been prescribed within two weeks of study enrollment.
* History of inhalational exposure (chemical, smoke, water, etc.) within 6 months of randomization
* Chest X-ray suggestive of granulomatous disease, malignancy, pneumonia, other acute pulmonary or pleural processes
* Current treatment with angiotensin converting enzyme (ACE) inhibitors
* Recent myocardial infarction, or history of congestive cardiac failure
* Active, concomitant disease which might limit the ability of the subject to participate in the study as determined by the Investigator (i.e., diabetes mellitus, congestive heart failure, unstable angina, etc.)
* Prior or current renal disease; calculated creatinine clearance < 30 mL/min (calculated CrCl < 30)
* History of Human Immunodeficiency Virus (HIV) or current clinically significant liver disease
* Use of opioids, neuromodulators (eg., gabapentin, pregabalin) first generation antihistamines (eg., diphenhydramine, chlorpheniramine) or antidepressants for the treatment of cough, during the study. Subjects taking drugs in these classes for chronic cough at time of screening may have them discontinued at least 2 days prior to randomization.
* Use of other NMDA-receptor antagonists (e.g. dextromethorphan, ketamine, amantadine) within 2 days of randomization
* Use of any of the following medications which may interact with memantine: quinidine, nicotine, neuroleptics such as chlorpromazine and promethazine, amitriptyline, baclofen, warfarin and hydrochlorothiazide
* Known hypersensitivity to memantine hydrochloride
* Observation of oral lesion(s) or abnormal finding(s) on oral cavity examination done at study screening or Day 0
* History of oropharyngeal leukoplakia, carcinoma or parotid dysfunction
* Subject has clinically significant abnormal laboratory test results at the screening visit (Subject may be enrolled by exception, as determined by the Principal Investigator and consented by Cerecor's Medical Monitor.)
* Subject has had clinically significant bleeding or donated blood or plasma within 30 days of randomization
* Subject has history of alcohol or drug abuse in past 2 years
* Subject has a positive drug and alcohol screen. Subjects receiving benzodiazepines by prescription, who test positive for benzodiazepines at the screening visit will be allowed.
* Subjects who have any disease or condition (medical or surgical) that might compromise hematologic, cardiovascular, pulmonary, renal, gastrointestinal, or central nervous system function; or any other conditions that might interfere with the absorption, distribution, metabolism, or excretion of the study drug, or that would place the subject at increased risk, as determined by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Cough Count/Frequency | Day 0-1, Day 14-15; Day 28-29, Day 42-43
  Change in start-to-end difference in cough count, active vs. placebo treatment periods

SECONDARY OUTCOMES:
LCQ | Days 0, 14, 28, & 42
  Start-to-end difference in Leicester Cough Questionnaire (LCQ) score, active vs. placebo treatment periods
VAS Score | Days 1, 14, 28, & 42
  Start-to-end difference in Visual analogue scale (VAS) score, active vs. placebo treatment periods
Cough Severity Diary | Days 0, 14, 28, & 42
  Start-to-end difference in CSD score, active vs. placebo treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Blake Paterson, MD, Study Chair — Avalo Therapeutics, Inc.
Locations (8):
- United States (8):
  - Allergy & Asthma Associates of Santa Clara Valley, San Jose, California
  - Sher Allergy Specialists, Largo, Florida
  - South Florida Clinical Research Trials, LLC, Miami, Florida
  - American Health Research, Charlotte, North Carolina
  - Wake Research, LLC, Raleigh, North Carolina
  - Oklahoma Institute of Allergy and Asthma, Oklahoma City, Oklahoma
  - Allergy, Asthma and Immunology Center, P.C./ Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Bellingham Asthma and Allergy Associates, Bellingham, Washington